CLINICAL TRIAL: NCT07221045
Title: PhytoRx Families: A Pilot Test Study to Address Food Security and Fruit and Vegetable Intake in Rural North Carolina
Brief Title: A Food As Medicine Approach to Address Food Insecurity in Rural North Carolina
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Collaborators: East Carolina University (Other)
Responsible Party: Principal Investigator, Basheerah Enahora, Assistant Professor, North Carolina State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 27407
Record Dates: First submitted 2025-10-20; First posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Diet, Healthy; Health Behavior; Blood Pressure; Diabetes Mellitus Risk; Utilization, Health Care
MeSH Terms: conditions — Health Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot test participants (Experimental): Participants will be referred by healthcare providers during office visits at local clinics. Providers will refer school-aged children (8-14 year olds) or adults, who are also a caregiver for a school-aged child, who screen positive for food insecurity and will submit patient referrals to the Project Coordinator utilizing a HIPAA-compliant KiteWorks platform.
  Interventions: Other: PhytoRx Families: A Pilot Test to Address Food Security in Rural North Carolina

INTERVENTIONS:
Other: PhytoRx Families: A Pilot Test to Address Food Security in Rural North Carolina — This project will pilot test and explore the impact of PhytoRx Families (PhtyoRxF) on nutrition-related, health-related, and healthcare utilization outcomes among n=30 adults and school-aged children (adult-child dyads; children 8-14 year olds, 2nd-9th grade).
  Other Names: PhytoRx Families Pilot Test

SUMMARY:
Increasing fruit and vegetable (FV) intake, and reducing saturated fat, salt, and added sugar are central lifestyle recommendations in the Dietary Guidelines for Americans to prevent chronic disease. Yet, while diet is modifiable, numerous barriers exist for lower-resourced families to engage in healthy dietary behaviors. In particular, rural families face structural and systemic disparities, such as inadequate access to affordable healthy food. Thus, this project. Thus, this study, PhytoRx Families, an innovative produce prescription (Prx) program, addresses health disparities in rural North Carolina (NC). This project will pilot test and explore the impact of PhytoRx Families (PhtyoRxF) on nutrition-related, health-related, and healthcare utilization outcomes.

DETAILED DESCRIPTION:
Increasing fruit and vegetable (FV) intake, and reducing saturated fat, salt, and added sugar are central lifestyle recommendations in the Dietary Guidelines for Americans to prevent chronic disease. Yet, while diet is modifiable, numerous barriers exist for lower-resourced families to engage in healthy dietary behaviors. In particular, rural families face structural and systemic inequities, such as inadequate access to affordable healthy food. Thus, this project, PhytoRx Families, an innovative produce prescription (Prx) program, will address health disparities in rural North Carolina (NC). This project will pilot test and explore the impact of PhytoRx Families (PhtyoRxF) on nutrition-related outcomes. This study will define impact on FV intake using the ASA24 dietary recall (primary outcome) among n=30 adults and school-aged children (adult-child dyads; children 8-14 year olds, 2nd-9th grade). The study will also explore the impact of PhytoRxF on cardiovascular health-related outcomes (blood pressure, glycated hemoglobin (HbA1C), height, weight (BMI calculated)). Finally the study will examine the change in healthcare utilization among PhytoRxF participants.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English or Spanish (speaking, reading, writing)
* An adult (18 years of age or older) who's a parent or caregiver of a child ages 8 to 14 years old or a child ages 8 to 14 years old
* Served at participating clinic in a county where the program is being implemented (Goldsboro Pediatrics, Bertie County Rural Health Association, and Roanoke Chowan Community Health in Bertie, Halifax, Lenoir, Northampton, or Wayne Counties)
* Living in a county where the program is being implemented (Bertie, Halifax, Lenoir, Northampton, or Wayne Counties)
* Free living to the extent they are able to receive and use a box of fresh produce and participate in direct nutrition education classes
* Willing and able to provide written consent and participate in all study activities.

Exclusion Criteria:

* Adults not at risk of food insecurity
* Adults, who are not parents nor caregivers of a child 8 to 14 years
* Adults who do not want to or could not fully participate (e.g., an adult family member with advanced kidney disease with severe dietary restrictions).

Ages: 8 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Fruit and vegetable intake | Baseline and end of study at 16 weeks
  Measured by ASA24 dietary recall

SECONDARY OUTCOMES:
Skin carotenoids | Baseline and end of study at 16 weeks
  Objective measure of fruit and vegetable intake measured by skin carotenoids, derived from a validated reflection spectroscopy device, Veggie Meter®
Diet quality | Baseline and end of study at 16 weeks
  Measured by ASA24 dietary recall
Food security status | Baseline and end of study at 16 weeks
  USDA 6-Item Food Security Survey. Score range is 0 to 6. Responses of "often" or "sometimes" on questions HH3 and HH4, and "yes" on AD1, AD2, and AD3 are coded as affirmative (yes). Responses of "almost every month" and "some months but not every month" on AD1a are coded as affirmative (yes). The sum of affirmative responses to the six questions in the module is the household's raw score on the scale. Food security status is assigned as follows: Raw score 0-1-High or marginal food security; Raw score 2-4-Low food security; Raw score 5-6-Very low food security
Nutrition security status | Baseline and end of study at 16 weeks
  4-Item Household Nutrition Security Screener (Gretchen Swanson/Center for Nutrition & Health Impact), Score range is 0 (if the participant selects "Always") to 4 (if the participant selects "Never"), with higher scores indicating a greater degree of Household Nutrition Security
Blood pressure | Baseline and end of study at 16 weeks
  Measured by automated monitor; Omron HEM-907XL, Vernon Hills
Hemoglobin A1C | Baseline and end of study at 16 weeks
  Measured by point-of-care (PoC) testing via A1C+ Now Analyzer, PTS Diagnostics
Body Mass Index | Baseline and end of study at 16 weeks
  Weight in kilograms and height in meters (collected at baseline only) will be assessed by electronic scale with stadiometer, SECA 874dr scale. BMI will be calculated by dividing weight (kg) by height (m) squared
Self-efficacy for Healthy Eating | Baseline and end of study at 16 weeks
  Self-efficacy for Eating Behaviors Scale. Score range from 1 (participant responds strongly disagree) to 5 (participant responds strongly agree), with higher scores indicating higher self efficacy for choosing healthy foods
Food-related Parenting Practices | Baseline and end of study at 16 weeks
  Comprehensive Home Environment Survey (CHES). Measurement of social and physical home environment to assess food-related parenting practices. Scale from 1 (participant responds "Never") to 5 (participant responds "Always"), with higher scores indicating positive food-related parenting practices (ie eating meals together as a family, modeling healthy behaviors, cooking at home, involving children in the meal planning/cooking process).
Barriers and Facilitators to Fruit and Vegetable Consumption | Baseline to end of study at 16 weeks
  Adapted instruments from the Family Life, Activity, Sun, Health, and Eating (FLASHE) Parent Module and the Singleton et al 2018 study to assess barriers and facilitators to fruit and vegetable consumption. Score range from 1 (participant responds "Strongly Disagree") to 5 (participant responds "Strongly Agree"), with higher scores representing more barriers to eating fruits and vegetables.
Body Mass Index-For-Age Percentile | Baseline and end of study at 16 weeks
  Weight in kilograms and height in meters (collected at baseline only) will be assessed by electronic scale with stadiometer, SECA 874dr scale. BMI will be calculated by dividing weight (kg) by height (m) squared, then plotted on a growth chart.

CONTACTS AND LOCATIONS:
Overall Officials: Basheerah Enahora, PhD, Principal Investigator — North Carolina State University
Locations (1):
- North Carolina State University, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data will be reported in aggregate for publication in academic journals (means and standard deviations). No identifying information will be reported in any publications arising from this research. No direct personal identifiers will be used in any published research.

REFERENCES:
- [Background] Norris K, Jilcott Pitts S, Reis H, Haynes-Maslow L. A Systematic Literature Review of Nutrition Interventions Implemented to Address Food Insecurity as a Social Determinant of Health. Nutrients. 2023 Aug 5;15(15):3464. doi: 10.3390/nu15153464. PMID 37571400
- [Background] Kerr D, Barua S, Glantz N, Conneely C, Kujan M, Bevier W, Larez A, Sabharwal A. Farming for life: impact of medical prescriptions for fresh vegetables on cardiometabolic health for adults with or at risk of type 2 diabetes in a predominantly Mexican-American population. BMJ Nutr Prev Health. 2020 Oct 5;3(2):239-246. doi: 10.1136/bmjnph-2020-000133. eCollection 2020 Dec. PMID 33521534
- [Background] Heasley C, Clayton B, Muileboom J, Schwanke A, Rathnayake S, Richter A, Little M. "I was eating more fruits and veggies than I have in years": a mixed methods evaluation of a fresh food prescription intervention. Arch Public Health. 2021 Jul 23;79:135. doi: 10.1186/s13690-021-00657-6. eCollection 2021. PMID 34301335
- [Background] Fischer L, Bodrick N, Mackey ER, McClenny A, Dazelle W, McCarron K, Mork T, Farmer N, Haemer M, Essel K. Feasibility of a Home-Delivery Produce Prescription Program to Address Food Insecurity and Diet Quality in Adults and Children. Nutrients. 2022 May 10;14(10):2006. doi: 10.3390/nu14102006. PMID 35631144
- [Background] Harkin N, Johnston E, Mathews T, Guo Y, Schwartzbard A, Berger J, Gianos E. Physicians' Dietary Knowledge, Attitudes, and Counseling Practices: The Experience of a Single Health Care Center at Changing the Landscape for Dietary Education. Am J Lifestyle Med. 2018 Nov 23;13(3):292-300. doi: 10.1177/1559827618809934. eCollection 2019 May-Jun. PMID 31105493
- [Background] Rahman V. Time to Revamp Nutrition Education for Physicians. Perm J. 2019;23:19-052. doi: 10.7812/TPP/19.052. Epub 2019 Aug 19. PMID 31496507
- [Background] Wolfson JA, Ramsing R, Richardson CR, Palmer A. Barriers to healthy food access: Associations with household income and cooking behavior. Prev Med Rep. 2019 Jan 31;13:298-305. doi: 10.1016/j.pmedr.2019.01.023. eCollection 2019 Mar. PMID 30792944
- [Background] Reicks M, Kocher M, Reeder J. Impact of Cooking and Home Food Preparation Interventions Among Adults: A Systematic Review (2011-2016). J Nutr Educ Behav. 2018 Feb;50(2):148-172.e1. doi: 10.1016/j.jneb.2017.08.004. Epub 2017 Sep 25. PMID 28958671
- [Background] Levi R, Schwartz M, Campbell E, Martin K, Seligman H. Nutrition standards for the charitable food system: challenges and opportunities. BMC Public Health. 2022 Mar 14;22(1):495. doi: 10.1186/s12889-022-12906-6. PMID 35287656
- [Background] Lutfiyya MN, Chang LF, Lipsky MS. A cross-sectional study of US rural adults' consumption of fruits and vegetables: do they consume at least five servings daily? BMC Public Health. 2012 Jun 1;12:280. doi: 10.1186/1471-2458-12-280. PMID 22490063
- [Background] Laraia BA. Food insecurity and chronic disease. Adv Nutr. 2013 Mar 1;4(2):203-12. doi: 10.3945/an.112.003277. PMID 23493536
- [Background] Backonja U, Park S, Kurre A, Yudelman H, Heindel S, Schultz M, Whitman G, Turner AM, Marchak NT, Bekemeier B. Supporting rural public health practice to address local-level social determinants of health across Northwest states: Development of an interactive visualization dashboard. J Biomed Inform. 2022 May;129:104051. doi: 10.1016/j.jbi.2022.104051. Epub 2022 Mar 19. PMID 35318149
- [Background] Byker Shanks C, Andress L, Hardison-Moody A, Jilcott Pitts S, Patton-Lopez M, Prewitt TE, Dupuis V, Wong K, Kirk-Epstein M, Engelhard E, Hake M, Osborne I, Hoff C, Haynes-Maslow L. Food Insecurity in the Rural United States: An Examination of Struggles and Coping Mechanisms to Feed a Family among Households with a Low-Income. Nutrients. 2022 Dec 9;14(24):5250. doi: 10.3390/nu14245250. PMID 36558409
- [Background] Schipper HS, de Ferranti S. Cardiovascular Risk Assessment and Management for Pediatricians. Pediatrics. 2022 Dec 1;150(6):e2022057957. doi: 10.1542/peds.2022-057957. PMID 36321395
- [Background] Harrington RA, Califf RM, Balamurugan A, Brown N, Benjamin RM, Braund WE, Hipp J, Konig M, Sanchez E, Joynt Maddox KE. Call to Action: Rural Health: A Presidential Advisory From the American Heart Association and American Stroke Association. Circulation. 2020 Mar 10;141(10):e615-e644. doi: 10.1161/CIR.0000000000000753. Epub 2020 Feb 10. PMID 32078375
- [Background] Abrahamowicz AA, Ebinger J, Whelton SP, Commodore-Mensah Y, Yang E. Racial and Ethnic Disparities in Hypertension: Barriers and Opportunities to Improve Blood Pressure Control. Curr Cardiol Rep. 2023 Jan;25(1):17-27. doi: 10.1007/s11886-022-01826-x. Epub 2023 Jan 9. PMID 36622491
- [Background] Ducharme-Smith K, Caulfield LE, Brady TM, Rosenstock S, Mueller NT, Garcia-Larsen V. Higher Diet Quality in African-American Adolescents Is Associated with Lower Odds of Metabolic Syndrome: Evidence from the NHANES. J Nutr. 2021 Jun 1;151(6):1609-1617. doi: 10.1093/jn/nxab027. PMID 33768240
- [Background] Esquivel Zuniga R, DeBoer MD. Prediabetes in Adolescents: Prevalence, Management and Diabetes Prevention Strategies. Diabetes Metab Syndr Obes. 2021 Nov 25;14:4609-4619. doi: 10.2147/DMSO.S284401. eCollection 2021. PMID 34858039
- [Background] Alberti KG, Zimmet P, Shaw J; IDF Epidemiology Task Force Consensus Group. The metabolic syndrome--a new worldwide definition. Lancet. 2005 Sep 24-30;366(9491):1059-62. doi: 10.1016/S0140-6736(05)67402-8. No abstract available. PMID 16182882
- [Background] Yang L, Magnussen CG, Yang L, Bovet P, Xi B. Elevated Blood Pressure in Childhood or Adolescence and Cardiovascular Outcomes in Adulthood: A Systematic Review. Hypertension. 2020 Apr;75(4):948-955. doi: 10.1161/HYPERTENSIONAHA.119.14168. Epub 2020 Mar 2. PMID 32114851
- [Background] Falkner B. The enigma of primary hypertension in childhood. Front Cardiovasc Med. 2022 Nov 4;9:1033628. doi: 10.3389/fcvm.2022.1033628. eCollection 2022. PMID 36407424